CLINICAL TRIAL: NCT01173055
Title: A Randomized, Double-blind,Placebo-controlled, Two-way Crossover Study to Evaluate the Effect of Milnacipran on Pain Processing and Functional Magnetic Resonance Imaging Activation Patterns in Patients With Fibromyalgia
Brief Title: A Study to Evaluate the Effects of Milnacipran on Pain Processing and Functional MRI in Patients With Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Daniel Clauw, MD, Daniel Clauw, Professor of Anesthesiology, University of Michigan, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MD-SAV-09
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milnacipran (Experimental): Milnacipran will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
  Interventions: Drug: milnacipran
- Placebo (Experimental): Placebo will be given orally twice daily in tablet form at different times during the course of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: milnacipran — Milnacipran will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
  Other Names: Savella
  Arms: Milnacipran
Drug: Placebo — Placebo will be given orally twice daily in tablet form at different times during the course of the study.
  Other Names: placebo/sugar pill
  Arms: Placebo

SUMMARY:
Fibromyalgia is a condition that includes pain, tenderness, stiff muscle, and fatigue. Researchers want to find out if "a drug" called milnacipran can help people with fibromyalgia. milnacipran (Savella) is approved by the FDA for the management of fibromyalgia. In this study, milnacipran will be given to find out more about how it affects pain and thinking in people with fibromyalgia.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effect of milnacipran on pain processing in patients with fibromyalgia and to assess the correlation between this effect and neural activation patterns during functional Magnetic Resonance Imaging (fMRI).

NOTE regarding Changes in Outcome Measures

In this Crossover Study, participants were involved for approximately 16 weeks in this sequence: a week of preparing for the initial assessments, baseline measurements (Week 0), 6 weeks on placebo or study drug followed by measurements for effect of drug or placebo (Week 6); a week of titration off of drug, if appropriate (or continued placebo, if on placebo), two weeks of washout, a new baseline assessment (Week 9), six weeks of study drug (or placebo), another set of measurements for effect of drug or placebo (Week 15), and a final titration period to maintain masking of assignment to drug or placebo. Of 17 participants who completed both sequences, data was analyzed for the 15 whose values for all measurement variables were usable.

When Outcome measure data was originally and accurately posted for baseline and change after treatment, the time frames listed were 0 and 15 weeks, because the last assessment was gathered at approximately week 15 for each person whose data is in the data set. However, given the crossover design, it seems more accurate and understandable, to show the time frame for the outcome measure as 6 because the participants were each administered drug or placebo for six weeks total. (Of course for the Placebo then Study Drug arm, the placebo data was collected at week 6, and for the Study Drug then Placebo arm, the drug data was collected at week 6, and similarly for the first group the drug data was collected at week 15 (first assignment, plus 1 week titration, 2 weeks washout, new baseline at week 9, and final collection at week 15), and for the second group the placebo data was collected at week 15.

Thus, outcome measures originally listed for 6 and 9 weeks, which were previously shown as "Data Not Reported" were effectively already included within the data presented for change from baseline shown in Week 15 in this fashion: 9 week data for the second assignment is part of the "week 0 data" for the first assignment, to get pre-treatment baseline for each treatment shown. Week 6 data is the post-treatment data which was shown as week 15, but is now recategorized as 6 week data. There is no, and never was, any data that could represent assignment to drug or placebo for 9 or 15 weeks.

Additionally, several outcome measures based on fMRI values were always listed in the protocol as other outcomes (not secondary outcomes), but had been incorrectly posted in the earlier listings on ClinicalTrials.gov. They have been accurately reclassified in the 2017 resubmission.

ELIGIBILITY:
Inclusion Criteria:

* You may be eligible to take part in this study if the following are true:

  * You are between the age of 18 and 70 years
  * If you are female
  * If you are right handed
  * You have a diagnosis of fibromyalgia for at least 3 months, as defined by the American College of Rheumatology 1990 Criteria
  * You are willing to stop taking certain medicines that you may be taking on a regular basis. The researchers will discuss these medications with you in detail

Exclusion Criteria:

* You may not be eligible take part in this study if any of the following are true for you:

  * You have problems with your heart or cardiovascular system
  * You have problems with your liver or kidneys
  * You have an autoimmune disease, or a whole-body infection like HIV or hepatitis
  * You have cancer
  * You are pregnant or breastfeeding
  * You abuse drugs or alcohol
  * You have suicidal thoughts or wishes
  * You have taken milnacipran or another study drug within the last 30 days
  * You have a medical problem not listed here that would make it unsafe for you to take part in the study
  * The research team feels that you will be unable to complete all phases of the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clauw, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Chronic Pain and Fatigue Research Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Ichesco E, Peltier SJ, Mawla I, Harper DE, Pauer L, Harte SE, Clauw DJ, Harris RE. Prediction of Differential Pharmacologic Response in Chronic Pain Using Functional Neuroimaging Biomarkers and a Support Vector Machine Algorithm: An Exploratory Study. Arthritis Rheumatol. 2021 Nov;73(11):2127-2137. doi: 10.1002/art.41781. Epub 2021 Sep 22. PMID 33982890

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants enrolled in the study received placebo for 1 week (Day -7 to 0) then began the double blinded treatment sequence.
Groups:
- Milnacipran First, Then Placebo: Milnacipran then placebo will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
  Milnacipran First, Then Placebo: Period 1 (Day 1-49); Milnacipran 12.5mg by mouth (PO) Day 1; 12.5mg twice daily (BID) Day 2 to 3; 25mg BID Day 4 to 7; 50mg BID Day 8-14; 100mg BID Day 15-42 followed by taper Day 43-49 and a 14 day washout period. Then, placebo matching study treatment in similar pattern to Period 1 was administered beginning Period 2 (Day 64-112).
- Placebo First, Then Milnacipran: Placebo, then milnacipran: Milnacipran and placebo will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
  Placebo First, Then Milnacipran: Period 1 (Day 1-49); Placebo matching study treatment was administered beginning Period 1 (Day 1-49) and a 14 day washout period. Then, Milnacipran Period 2 (Day 64-112); Milnacipran 12.5mg Day 62; 12.5mg twice daily (BID) Day 65 to 66; 25mg BID Day 67 to 70; 50mg BID Day 71-77; 100mg BID Day 78-105 followed by taper Day 106-112.
Period: Period 1 - Day 1 to 49
Arm/Group | Milnacipran First, Then Placebo | Placebo First, Then Milnacipran
Started | 10 | 12
Completed | 8 | 10
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Placebo Washout Period - Day 50 to 63
Arm/Group | Milnacipran First, Then Placebo | Placebo First, Then Milnacipran
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0
Period: Period 2 - Day 64 to 112
Arm/Group | Milnacipran First, Then Placebo | Placebo First, Then Milnacipran
Started | 8 | 10
Completed | 8 | 9
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: The milnacipran then placebo arm was reduced from eight to six participants for the analysis due to tolerating a dose of Milnacipran less than 200mg/day. This was done to be consistent with the dosing of all other participants.
Groups:
- Milnacipran First, Then Placebo: Milnacipran and placebo will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
  milnacipran, then placebo: Milnacipran and placebo will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
- Placebo First, Then Milnacipran: Milnacipran and placebo will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
  Placebo, then milnacipran: Milnacipran and placebo will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
- Total: Total of all reporting groups
Arm/Group | Milnacipran First, Then Placebo | Placebo First, Then Milnacipran | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Customized [Mean (Standard Deviation); unit: years]
  Fibromyalgia | 46.83 (9.83) | 36.67 (8.64) | 40.73 (10.187)
Sex/Gender, Customized [Number; unit: participants]
  Female | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pain Threshold at Baseline
Description: The primary outcome parameter is the medium pressure pain threshold at pre-treatment baseline (pressure that evokes a perceived pain intensity of 40-50 out of 100 on a numerical rating scale). Measured in kg/cm^2.
Time Frame: Baselines measured at week 0 and week 9 after washout from first assignment to treatment
Measure: Mean (Standard Deviation); unit: kg/cm^2
Groups:
- Milnacipran: Milnacipran and placebo will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
  milnacipran, then placebo: Milnacipran and placebo will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
- Placebo: Milnacipran and placebo will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
  Placebo, then milnacipran: Milnacipran and placebo will be given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
kg/cm^2 | 2.7333 (.83166) | 2.583 (.84339)

2. Primary Outcome: Change in Pain Threshold From Baseline to End of Treatment.
Description: The primary outcome parameter is the change in medium pressure pain threshold (pressure that evokes a perceived pain intensity of 40-50 out of 100 on a numerical rating scale) from baseline to end of treatment. Measured in kg/cm^2. Lower values represent a worse outcome.
Time Frame: baseline compared with 6 weeks of treatment
Population: Of 17 participants who completed both sequences, data was analyzed for the 15 whose values for all measurement variables were usable.
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
kg/cm^2
  Pre-Treatment (Week 0 or 9) | 2.7333 (.83166) | 2.583 (.84339)
  Post-Treatment (Week 6 or 15) | 2.650 (1.05982) | 2.70 (.99642)

3. Secondary Outcome: Diffuse Noxious Inhibitory Control (DNIC) Effect at Baseline.
Description: 0-100 numerical rating scale. 0 on the numerical scale represents a better outcome. 100 represents a worse outcome.
Time Frame: Baselines measured at week 0 and week 9 after washout from first assignment to treatment
Population: One participant did not complete this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 14
units on a scale | 8.134 (17.51978) | 12.0240 (20.80824)

4. Secondary Outcome: Change in Diffuse Noxious Inhibitory Control (DNIC) Effect From Baseline to End of Treatment.
Description: 0-100 numerical rating scale. 0 on the numerical scale represents a better outcome. 100 represents a worse outcome.
Time Frame: baseline compared with 6 weeks of treatment
Population: Of 17 participants who completed both sequences, data was analyzed for the 15 whose values for all measurement variables were usable. On the placebo, side one additional participant did not have data for this variable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 14
units on a scale
  Pre-Treatment (Week 0 or 9) | 8.134 (17.51978) | 12.0240 (20.80824)
  Post-Treatment (Week 6 or 15) | 11.0355 (17.16822) | 8.50 (19.6678)

5. Secondary Outcome: Pain Tolerance at Baseline
Description: The primary outcome parameter is the pressure pain tolerance (maximum tolerated pressure) at pre-treatment baseline.
Time Frame: Baselines measured at week 0 and week 9 after washout from first assignment to treatment
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
kg/cm^2 | 4.2667 (1.39983) | 3.80 (1.17716)

6. Secondary Outcome: Change in Pain Tolerance From Baseline to End of Treatment
Description: The primary outcome parameter is the change in pressure pain tolerance (maximum tolerated pressure) from baseline to end of treatment. Measured in kg/cm^2. Lower values represent a worse outcome.
Time Frame: baseline compared wtih 6 weeks of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 15 | 15
kg/cm^2
  Pre-Treatment (Week 0 or 9) | 4.2667 (1.39983) | 3.80 (1.17716)
  Post-Treatment (Week 6 or 15) | 3.8667 (1.43261) | 3.8667 (1.20218)

7. Other Pre Specified Outcome: Change in fMRI Brain Activation Patterns During Pressure Stimulation From Baseline to End of Treatment
Time Frame: Baselines measured at week 0 and week 9 after washout from first assignment to treatment; treatment effect measures collected 6 weeks later
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Descending Pain Modulation From Baseline to End of Treatment (as Assessed by Changes in fMRI Brainstem Activation Patterns)
Time Frame: as for outcome 7
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in fMRI Activation Patterns During N-back Procedure From Baseline to End of Treatment.
Time Frame: as for outcome 7
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Milnacipran: Milnacipran was given orally twice daily in tablet form at different times during the course of the study. The highest dose of milnacipran to be used in the study is 200mg/day.
- Placebo: Placebo was given orally twice daily in tablet form at different times during the course of the study.
Arm/Group | Milnacipran | Placebo
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 13/20 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=20) | Placebo (N=20)
Herniated Disc (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=20) | Placebo (N=20)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 4 (4)
Distrubance in Attention (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Increased Blood Pressure (Cardiac disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hot Flashes (Vascular disorders) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Sensitive to Light (Eye disorders) | 1 (1) | 0 (0)
Sore Eyes (Eye disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 2 (3) | 2 (2)
Emotional (Psychiatric disorders) | 1 (1) | 1 (1)
Food Poisioning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough/Congestion (Infections and infestations) | 1 (1) | 0 (0)
Unable to Void (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Raw Tongue (General disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less